CLINICAL TRIAL: NCT00139672
Title: A Multi-Center, Double-Blind, Randomized, Placebo-Controlled, Parallel Group Study To Investigate The Effect Of Pd-217,014 In Patients With Irritable Bowel Syndrome (IBS)
Brief Title: A Study To Investigate The Effect Of PD-217,014 On Abdominal Pain/Discomfort In Patients With IBS.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A4451007
Record Dates: First submitted 2005-08-29; First posted 2005-08-31 (Estimated); Last update posted 2008-06-17 (Estimated); Status verified 2008-06

CONDITIONS: Irritable Bowel Syndrome
MeSH Terms: conditions — Irritable Bowel Syndrome

INTERVENTIONS:
Drug: PD-217,014

SUMMARY:
The purpose of this study is to determine the effectiveness of PD-217,014 in the treatment of abdominal pain/discomfort associated with irritable bowel disease.

ELIGIBILITY:
Inclusion Criteria:

* Males and females having Irritable bowel syndrome as defined by the Rome II criteria.
* Patients must have had normal examination of colon anatomy within the last 5 years

Exclusion Criteria:

* Patient with an organic gastrointestinal disease.
* Patients with poor renal function.
* Patients with severe constipation.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 330
Dates: Start 2004-01; Primary Completion 2005-02 (Actual); Study Completion 2005-02 (Actual)

PRIMARY OUTCOMES:
Assess the effect of PD-217,014 on the relief of abdominal pain/discomfort in patients with irritable bowel syndrome. Primary endpoint is a responder, defined by having adequate relief for > or = 50% of the active treatment period (4 weeks).

SECONDARY OUTCOMES:
Assess the effect of PD-217,014 on the patient's global assessment of IBS symptoms, stool frequency & consistency and on abdominal bloating (change from baseline to week 4).

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer